CLINICAL TRIAL: NCT05589727
Title: Study to Validate the Application of the Epidemiological Diagnostic Criteria of Ventilator-Associated Events (VAE) in Ventilator-Associated Pneumonia (VAP) Notified to the Brazilian Health Regulatory Agency (ANVISA)
Brief Title: Application of Ventilator-Associated Events (VAE) in Ventilator-Associated Pneumonia (VAP) Notified in Brazil
Status: Completed | Type: Observational
Sponsor: Giovanna Marssola Nascimento (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor-Investigator, Giovanna Marssola Nascimento, Principal Investigator, Hospital Alemão Oswaldo Cruz
Organization: Hospital Alemão Oswaldo Cruz (Other)
Other Study IDs: IMPACTO MR-PAV
Record Dates: First submitted 2022-10-13; First posted 2022-10-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Ventilator-Associated Pneumonia; Healthcare-Associated Pneumonia; Healthcare Associated Infection
Keywords: pneumonia; surveillance; healthcare associated infections; Ventilator-Associated Pneumonia; Healthcare-Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Cross Infection; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with VAP - ANVISA criteria: Patients notified with Ventilator-Associated Pneumonia (VAP) when using the current ANVISA criteria.
- Patients with VAP - NHSN criteria: Patients notified with Ventilator-Associated Pneumonia (VAP) when using the Ventilator-Associated Events (VAE) criteria defined by the NHSN.

SUMMARY:
Multicentric observational prospective cohort study in 12 (twelve) hospitals representing all Brazilian regions.

The main objective of this project is to evaluate the incidence of Ventilator-Associated Pneumonia (VAP) when using the current ANVISA criteria for VAP versus VAE criteria defined by the National Healthcare Safety Network (NHSN). The diagnostic accuracy of the two criteria for identifying VAP will also be compared, characterizing other events associated with mechanical ventilation that are not VAP, when applicable.

The study also aims to adjudicate ventilator-associated pneumonias reported to ANVISA using current epidemiological diagnostic criteria.

DETAILED DESCRIPTION:
The study will be carried out in about 12 centers, comprising the five Brazilian regions. It will be conducted from 2022 to 2024. Data collection will be performed at each center during six months.

Trained health professionals from Infections Control Committees of each participating center will collect data.

Mechanical ventilation data will be entered daily in the database system from the moment the patient is submitted to mechanical ventilation until the first day after the end of mechanical ventilation.

VAPs notified to ANVISA, according to its own criteria, will be reported monthly in the database system for adjudication.

The VAE definition will be performed automatically in the database system by mans of a specific algorithm. The diagnosis established by the system will be manually validated by a nurse with experience in healthcare-associated infection (HAI) surveillance. Agreement variables (Kappa) between the two criteria will be analyzed.

The adjudication will be carried out by two independent professionals (doctor and nurse) with experience in HAIs surveillance. In case of disagreement, there will be an evaluation by a third adjudicator.

The complete project was submitted to the local Institutional Review Board (IRB)/National Research Ethics Commission (CONEP) system and has ethical approval (CAAE: 52354721.0.1001.0070).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Pacients hospitalized in intensive care units (ICUs) using mechanical ventilation

Exclusion Criteria:

* Patients withdrawn from mechanical ventilation (MV) on the first day (D1) or second day (D2), with D1 being the day of initiation of MV;
* Patients with hospital discharge (discharge, death or transfer) on D1 or D2 of mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years or older who are hospitalized in intensive care units (ICUs) using mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 987 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Ventilator-Associated Pneumonia (VAP) using two different surveillance criteria. | through study completion, an average of 6 months
  To evaluate the incidence of Ventilator-Associated Pneumonia (VAP) when using the current ANVISA criteria for VAP versus the criteria for events Ventilator-Associated Events (VAE) defined by the NHSN.

SECONDARY OUTCOMES:
Accuracy of the two criteria for identifying VAP | through study completion, an average of 6 months
  The diagnostic accuracy of the two criteria for identifying VAP will also be compared, characterizing other events associated with mechanical ventilation other than VAP, when applicable - Ventilator-Associated Condition (VAC), Infection-related Ventilator-Associated Complication (IVAC), Possible Ventilator-Associated Pneumonia (PVAP).
Adjudication of VAP | through study completion, an average of 6 months
  To adjudicate ventilator-associated pneumonias reported to ANVISA using current epidemiological diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna M Nascimento, MD, Principal Investigator — Hospital Alemão Oswaldo Cruz
Locations (12):
- Brazil (12):
  - Hospital São Vicente de Paula, Barbalha, Ceará
  - Hospital OTOclínica, Fortaleza, Ceará
  - Hospital Universitário de Brasília, Brasília, Federal District
  - Hospital Geral de Goiânia Alberto Rassi, Goiânia, Goiás
  - Hospital Presidente Vargas, São Luís, Maranhão
  - Hospital Municipal de Maringá, Maringá, Paraná
  - Hospital Jean Bittar, Belém, Pará
  - Hospital do Tricentenário, Olinda, Pernambuco
  - Instituto Estadual do Cérebro Paulo Niemeyer, Rio de Janeiro, Rio de Janeiro
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Do Grande Do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - A. C. Camargo Cancer Center, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Klompas M. Ventilator-Associated Events: What They Are and What They Are Not. Respir Care. 2019 Aug;64(8):953-961. doi: 10.4187/respcare.07059. PMID 31346070
- [Background] Klompas M. The paradox of ventilator-associated pneumonia prevention measures. Crit Care. 2009;13(5):315. doi: 10.1186/cc8036. Epub 2009 Oct 15. PMID 19849825
- [Background] Fan Y, Gao F, Wu Y, Zhang J, Zhu M, Xiong L. Does ventilator-associated event surveillance detect ventilator-associated pneumonia in intensive care units? A systematic review and meta-analysis. Crit Care. 2016 Oct 24;20(1):338. doi: 10.1186/s13054-016-1506-z. PMID 27772529
- [Background] Raoof S, Baumann MH; Critical Care Societies Collaborative, consisting of the leadership of the American Association of Critical-Care Nurses, the American College of Chest Physicians, the American Thoracic Society, and the Society of Critical Care Medicine. Ventilator-associated events: the new definition. Am J Crit Care. 2014 Jan;23(1):7-9. doi: 10.4037/ajcc2014469. No abstract available. PMID 24382609
- [Background] Stevens JP, Silva G, Gillis J, Novack V, Talmor D, Klompas M, Howell MD. Automated surveillance for ventilator-associated events. Chest. 2014 Dec;146(6):1612-1618. doi: 10.1378/chest.13-2255. PMID 25451350
- [Background] Hebert C, Flaherty J, Smyer J, Ding J, Mangino JE. Development and validation of an automated ventilator-associated event electronic surveillance system: A report of a successful implementation. Am J Infect Control. 2018 Mar;46(3):316-321. doi: 10.1016/j.ajic.2017.09.006. Epub 2017 Nov 10. PMID 29132696
- [Background] Sim J, Wright CC. The kappa statistic in reliability studies: use, interpretation, and sample size requirements. Phys Ther. 2005 Mar;85(3):257-68. PMID 15733050
- [Background] Donner A, Eliasziw M. A goodness-of-fit approach to inference procedures for the kappa statistic: confidence interval construction, significance-testing and sample size estimation. Stat Med. 1992 Aug;11(11):1511-9. doi: 10.1002/sim.4780111109. PMID 1410963
- [Derived] Nascimento GM, Rodrigues DLG, Piastrelli FT, Cheno MY, Braz KCC, Alves LBO, Tomazini BM, Veiga VC, Arns B, Besen BAMP, Junior APN, Avezum A, da Silva RKL, de Azevedo CMPES, Silva MLSO, Kist GR, Salgado FB, de Moura MTF, Boschi E, Kurtz PMP, Miraglia ERVDS, de Lima TA, Pereira RR, Arraes JA, Alves de Oliveira Junior H. Ventilator-associated events criteria in the assessment of Ventilator-Associated Pneumonia (IMPACTO MR-PAV): A prospective cohort. Braz J Infect Dis. 2025 Jul-Aug;29(4):104543. doi: 10.1016/j.bjid.2025.104543. Epub 2025 May 22. PMID 40409133
- [Derived] Nascimento GM, Gomes Rodrigues DL, Mangas Catarino DG, Piastrelli FT, Cheno MY, Braz KCC, Oliveira Alves LB, Avezum A, Veiga VC, Zavascki AP, Tomazini B, Besen B, Pereira AJ, Marques de Pinho APN, De Oliveira Junior HA. Application of ventilator-associated events (VAE) in ventilator-associated pneumonia (VAP) notified in Brazil (IMPACTO MR-PAV): a protocol for a cohort study. BMJ Open. 2023 Dec 9;13(12):e076047. doi: 10.1136/bmjopen-2023-076047. PMID 38070904